CLINICAL TRIAL: NCT04754776
Title: A Phase I Study to Determine the Safety & Immunogenicity of the Candidate Rift Valley Fever Virus (RVFV) Vaccine ChAdOx1 RVF in UK Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity of a Candidate RVFV Vaccine (RVF001)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RVF001
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-04

CONDITIONS: Rift Valley Fever
Keywords: RVF; ChAdOx1; vaccine
MeSH Terms: conditions — Rift Valley Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): 5 x 10^9 vp ChAdOx1 RVF delivered intramuscularly
  Interventions: Biological: ChAdOx1 RVF
- Medium dose (Experimental): 2.5 x 10^10 vp ChAdOx1 RVF delivered intramuscularly
  Interventions: Biological: ChAdOx1 RVF
- High dose (Experimental): 5 x 10^10 vp ChAdOx1 RVF delivered intramuscularly
  Interventions: Biological: ChAdOx1 RVF

INTERVENTIONS:
Biological: ChAdOx1 RVF — Single dose of ChAdOx1 RVF

SUMMARY:
Phase I open label, non-randomised dose escalation study on healthy UK volunteers aged from 18 to 50 years to assess the safety and immunogenicity of ChAdOx1 RVF

DETAILED DESCRIPTION:
The purpose of this study is to test a new vaccine against the Rift Valley Fever Virus (RVFV) in healthy volunteers.

Rift Valley fever is a disease caused by RVFV and it is transmitted to humans through a mosquito bite or contact with virus-contaminated tissues and fluids. Although initially restricted to Africa, the virus can be transmitted by several different mosquito species that are more widely distributed than the virus itself, leading to concerns of disease spread as has occurred in the Arabian Peninsula and Madagascar. In humans, RVFV infection usually presents as a sudden febrile illness, but severe manifestations including bleeding disorders and neurological complications may also occur. RVFV is considered a global health threat with significant potential for international spread and use in bioterrorism.

Vaccines against RVFV are available for livestock, however no licensed vaccines or specific treatments are currently available for humans.

The study will enable assessment of the safety of the new vaccine called ChAdOx1 RVF and the extent of immune response in healthy volunteers. Healthy adult volunteers will receive a single dose of a new candidate vaccine at different doses. The objective of this first-in-human study is to find the optimal dose of the vaccine, balancing immune responses and profile of adverse events.

Healthy volunteers aged 18-50 will be recruited in Oxford and vaccinated at the Centre for Clinical Vaccinology and Tropical Medicine and will be followed for a period of 3 months. The study is funded by the UK Biotechnology and Biological Sciences Research Council(BBSRC) and the Medical Research Council (MRC)/Department of Health, through the UK Vaccines Network.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

1. Healthy adults aged 18 to 50 years
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner or access this medical history electronically
4. For females only, willingness to practice continuous effective contraception for at least 3 months and a negative pregnancy test on the day(s) of screening and vaccination
5. Agreement to refrain from blood donation during the course of the study
6. Able to provide written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data.
3. Prior receipt of any vaccines administered ≤30 days before enrolment and/or planned receipt of a vaccine ≤30 days after enrolment EXCEPT for protein, RNA (or other non-adenovirus based) COVID-19 vaccinations which may be given within 14 days of the trial vaccine.
4. Receipt of a recombinant simian adenoviral vaccine prior to enrolment
5. Planned receipt of another adenoviral vectored vaccine (e.g. Oxford/Astrazeneca or Janssen COVID-19 vaccines) within 90 days after the vaccination with the ChAdOx1 RVF
6. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
7. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
8. COVID-19 infection diagnosed in the community in the 28 days prior to enrolment
9. Any main covid-19 symptom within 28 days of enrolment:

   1. Fever (subjective or ≥37.8)
   2. New continuous cough
   3. Loss of sense of smell
   4. Loss of sense of taste
10. Clinical suspicion of acute COVID-19 in the 28 days prior to enrolment
11. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
12. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
13. Any history of anaphylaxis in relation to vaccination
14. Pregnancy, lactation or willingness/intention to become pregnant during the study
15. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
16. History of serious psychiatric condition likely to affect participation in the study
17. Bleeding disorder (eg. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
18. Any other serious chronic illness requiring hospital specialist supervision
19. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
20. Suspected or known injecting drug abuse in the 5 years preceding enrolment
21. Seropositive for hepatitis B surface antigen (HBsAg)
22. Seropositive for hepatitis C virus (antibodies to HCV)
23. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
24. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
25. Inability of the study team to contact the volunteer's GP (or access summary care record, if available) to confirm medical history and safety to participate
26. Prior natural exposure to RVFV as determined by seropositivity for RVFV antigens by ELISA and neutralizing antibody assay (serology will be requested at the discretion of the investigator)
27. History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism), history of antiphospholipid syndrome, or history of heparin induced thrombocytopenia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
To assess local reactogenicity | 7 days following vaccination
  Occurrence of solicited local reactogenicity signs and symptoms
To assess systemic reactogenicity | 7 days following vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms
To assess unsolicited adverse events | 28 days following vaccination
  Occurrence of unsolicited adverse events
To assess the safety and tolerability of ChAdOx1 RVF in healthy adult volunteers | Duration of study (6 months)
  Frequency of participants with clinically significant changes from baseline safety laboratory measures (haematology and biochemistry blood results)
To assess serious adverse events | Duration of study (6 months)
  Occurrence of serious adverse events

SECONDARY OUTCOMES:
Assess the cellular and humoral immunogenicity of ChAdOx1 RVF in healthy adult volunteers | Duration of study (6 months)
  ELISA to quantify antibodies to GnGc proteins
Assess the cellular and humoral immunogenicity of ChAdOx1 RVF in healthy adult volunteers | Duration of study (6 months)
  RVFV neutralising antibody titres
Assess the cellular and humoral immunogenicity of ChAdOx1 RVF in healthy adult volunteers | Duration of study (6 months)
  Ex vivo ELISpot and flow cytometry responses to GnGc

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Prof, Principal Investigator — Jenner Institute
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkin D, Wright D, Folegatti PM, Platt A, Poulton I, Lawrie A, Tran N, Boyd A, Turner C, Gitonga JN, Karanja HK, Mugo D, Ewer KJ, Bowden TA, Gilbert SC, Charleston B, Kaleebu P, Hill AVS, Warimwe GM. Safety and immunogenicity of a ChAdOx1 vaccine against Rift Valley fever in UK adults: an open-label, non-randomised, first-in-human phase 1 clinical trial. Lancet Infect Dis. 2023 Aug;23(8):956-964. doi: 10.1016/S1473-3099(23)00068-3. Epub 2023 Apr 13. PMID 37060917

DOCUMENTS (1):
  • Study Protocol (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04754776/Prot_000.pdf